CLINICAL TRIAL: NCT06641310
Title: Phase 1a/b Trial of Exercise Therapy in Familial Adenomatous Polyp (FAP)
Brief Title: Trial of Exercise Therapy in Familial Adenomatous Polyp (FAP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UMCC 2024.083; NCI-2023-10925 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00256140 (Other: University of Michigan Rogel Cancer Center); UMI23-15-01 (Other: DCP); UG1CA242632 (NIH)
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Familial Adenomatous Polyposis
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise therapy comprising treadmill walking (Experimental): exercise therapy
  Interventions: Procedure: Exercise Therapy

INTERVENTIONS:
Procedure: Exercise Therapy — Exercise therapy comprising treadmill walking will be administer by exercise physiologists via a study-kit which includes a smart-watch (activity tracker), heart rate monitor, blood pressure cuff, body composition scale, and e-tablet for remotely monitoring your exercise. The trials will test 3 exercise levels (150, 225, and 300 minutes per week), with one de-escalation exercise level of 90 minutes per week if needed.

SUMMARY:
The purpose of this phase 1a/b trial is to find out what amount of exercise would be best to use for preventing recurrence of colorectal polyps. It involves following one of four different amounts of exercise regimens on a treadmill for 26 weeks. A treadmill will be placed in each study participant's home for the duration of the study. The exercise regimen will be personalized for each participant and monitored remotely by exercise personnel. The in-person study visits occur during the usual standard of care endoscopy exam and during a follow-up exam that is 26 weeks later. Small rectal tissue biopsies, about the size of a grain of rice, will be taken before and after 26 weeks of exercise. The study visits also involve questionnaires, a stool sample, and a blood sample. This study will inform the design of larger, future trials to investigate whether or not recurrence of polyps can be achieved with exercise.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with FAP as defined by:

  * Genetic diagnosis: APC germline mutation (with or without FAP family history), OR
  * Clinical diagnosis: FAP phenotype with a history of more than 50 colorectal adenomas
* Have an intact rectum defined as status post colectomy and ileocolonic anastomosis for polyposis or pre-colectomy
* ≥ 5 rectal polyps > 2 mm in size on baseline lower endoscopy
* Participants must have no evidence of invasive cancer for 6 months prior to screening and must be at least 6 months from any prior cancer-directed treatment (such as surgical resection, chemotherapy, immunotherapy, hormonal therapy or radiation)
* No initiation of daily use of sulindac, celecoxib or other non-steroidal anti-inflammatory medications (NSAIDs) within 3 months of day 1 and no initiation > 25% of the time (> 8 days/month) for the duration of study participation
* No initiation of semaglutide, liraglutide (glucagon-like peptide-1 receptor agonist [GLP-1 receptor agonist]), tirzepatide (glucose-dependent insulinotropic polypeptide [GIP]), orlistat (lipase inhibitor) or other weight loss medications, within 3 months of day 1 and during study participation
* Adults ≥ 18 years of age
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Participants on chronic suppressive antiviral therapy for herpes simplex virus (HSV) are eligible
* Lower endoscopy, required for participation in the study, is contraindicated in pregnancy. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation, and until after the end of study endoscopy is completed. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform the study team immediately
* Inactive defined as ≤ 60 minutes of moderate or strenuous exercise per week over the past month as assessed by the Godin Leisure Time Exercise Questionnaire
* No self-reported contraindications to regular exercise as evaluated by the Physical Activity Readiness Questionnaire (PAR-Q+)
* Sufficient space to house a treadmill in primary residence for the intervention period or access to an approved treadmill (as determined by study exercise physiologist) for the intervention period (e.g., participant may have access to a treadmill via an existing membership to a health club)
* Ability for study team to deliver and install exercise equipment in primary residence

  * Note: If participant will be using treadmill from another source approved by study exercise physiologist, this inclusion criteria is not applicable
* Internet or Wi-Fi connection. For participants without internet or Wi-Fi, a pre-paid cellular iPad will be provided
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Physician approval
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* History of total proctocolectomy
* Histologically-confirmed high-grade dysplasia or cancer on biopsy at screening
* History of pelvic radiation
* Participants receiving any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of severe, progressive, or uncontrolled renal, genitourinary, hepatic, hematologic, endocrine, cardiac, vascular, pulmonary, rheumatologic, neurologic, psychiatric, or metabolic disturbances, or signs and symptoms thereof
* Pregnant women are excluded since endoscopy is not recommended while pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Exercise therapy compliance (feasibility) | between 4-12 weeks
  Compliance to the planned treatment regimen will be evaluated by the ratio of completed versus planned level of exercise therapy at each level tested.

SECONDARY OUTCOMES:
Physiological changes | Baseline up to 26 weeks
  Exercise capacity will be evaluated by a sub-maximal exercise capacity test.

OTHER OUTCOMES:
Change in the proliferation and apoptosis | up to 27 weeks
  To evaluate change in the proliferation and apoptosis in rectal adenomas and normal appearing rectal mucosa from baseline to end of treatment
Change in the proliferation / apoptosis ratio | up to 27 weeks
  To evaluate change in the proliferation / apoptosis ratio in rectal adenomas and normal appearing rectal mucosa from baseline to end of treatment
Change in rectal polyp burden | up to 27 weeks
  To evaluate the change in rectal polyp burden from baseline to end of treatment
Changes in body composition | up to 27 weeks
  To evaluate physiological response to exercise therapy as evaluated by changes in body composition
Changes in lifestyle | up to 27 weeks
  To evaluate changes in lifestyle states (general physical activity performed outside of structured and diet) during intervention with exercise therapy

CONTACTS AND LOCATIONS:
Overall Officials: Samara Rifkin, MD, Principal Investigator — University of Michigan Rogel Cancer Center; Lee Jones, Ph.D, Principal Investigator — City of Hope Medical Center; Carol Burke, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Cleveland Clinic Foundation, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared